CLINICAL TRIAL: NCT04615455
Title: A Randomized Clinical Trial Evaluating Allogeneic Adipose-derived MesenchymAl Stem Cells as a Treatment of Dry Eye Disease in Patients With Sjögren's Syndrome
Brief Title: Mesenchymal Stem Cell Therapy of Dry Eye Disease in Patients With Sjögren's Syndrome
Acronym: AMASS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Møller-Hansen, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-002804-38
Record Dates: First submitted 2020-11-03; First posted 2020-11-04 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Keratoconjunctivitis Sicca, in Sjogren's Syndrome
MeSH Terms: conditions — Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adipose tissue-derived mesenchymal stem cells (ASCs) (Experimental): One transconjunctival injection of allogeneic ASCs into the LG in one eye.
  Interventions: Drug: ASCs
- Placebo (vehicle, Cryostor CS10) (Placebo Comparator): One transconjunctival injection of Cryostor CS10 into the LG in one eye.
  Interventions: Drug: Cryostor CS10

INTERVENTIONS:
Drug: ASCs — ASCs expanded from healthy donors. The ASC product contains 22 million ASCs/ml.
  Other Names: Allogeneic adipose-derived mesenchymal stem cells
  Arms: Adipose tissue-derived mesenchymal stem cells (ASCs)
Drug: Cryostor CS10 — CryoStor® CS10 freeze medium
  Arms: Placebo (vehicle, Cryostor CS10)

SUMMARY:
AMASS is a double-blinded randomized clinical trial with the purpose of investigating whether injection of allogeneic adipose-derived mesenchymal stem cells (ASCs) into the lacrimal gland (LG) results in increased ocular comfort compared to placebo.

DETAILED DESCRIPTION:
AMASS is a double-blinded randomized clinical trial which will be performed at the Department of Ophthalmology, University Hospital of Copenhagen, Denmark. 40 patients with severe aqueous deficient dry eye disease (ADDE) due to Sjögren's Syndrome (SS) will be recruited from the Dept. of Ophthalmology, Rigshospitalet, and allocated in ratio 1:1 to either injection of allogeneic adipose-derived mesenchymal stem cells (ASCs) or placebo (vehicle, Crystore CS10) into the lacrimal gland (LG) in one eye. We hypothesize that injection of allogeneic ASCs into the LG increases tear production and reduce inflammation resulting in increased ocular comfort compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sjögren's syndrome according to the 2016 American College of Rheumatology/European League Against Rheumatism classification criteria for primary Sjögren's syndrome
* OSDI-score ≥ 33
* Schirmer's test 1-5 mm/5 minutes
* NIKBUT < 10 sec

Exclusion Criteria:

* LG volume on MRI < 0,2 cm3 in the study eye
* Previous treatment with ASCs or other stem cell products in the LG(s)
* Reduced immune response (e.g. HIV positive)
* Pregnancy or planned pregnancy within the next 2 years
* Breastfeeding
* Topical treatment with eye drops other than to treat dry eye disease (DED)
* Any other disease/condition judged by the investigator to be grounds for exclusion, such as infection in or around the eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | 4 months after treatment
  The OSDI is a valid and reliable instrument for measuring dry eye disease severity

SECONDARY OUTCOMES:
Non-invasive keratography tear break-up time (NIKBUT) | 4 months after treatment
  As measured with the Keratograph 5M (Oculus™)
Tear meniscus height (TMH) | 4 months after treatment
  As measured with the Keratograph 5M (Oculus™)
Schirmer's I test | 4 months after treatment
  Change in tear production as evaluated with the Schirmer's I test
Tear osmolarity | 4 months after treatment
  Change in tear osmolarity measured with TearLab™
Oxford scale | 4 months after treatment
  Change in staining of the ocular surface (grade 0-5 with 0 being absent corneal staining and 5 being severe corneal staining)
HLA anti-bodies | 12 months after treatment
  Development of anti-human leucocyte antigen (HLA) anti-bodies evaluated with Luminex HLA anti-body screening
  Development of anti-HLA anti-bodies evaluated with Luminex HLA anti-body screening
  Development of donor-specific HLA-antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Heegaard, MD, DMSc, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, DK, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen AC, Moller-Hansen M, Wiencke AK, Terslev L, Torp-Pedersen S, Heegaard S. Ultrasound-Guided Transcutaneous Injection in the Lacrimal Gland: A Description of Sonoanatomy and Technique. J Ocul Pharmacol Ther. 2023 May;39(4):275-278. doi: 10.1089/jop.2022.0156. Epub 2023 Mar 21. PMID 36944128